CLINICAL TRIAL: NCT00003821
Title: Phase II Trial of Aminopterin in Patients With Persistent or Recurrent Endometrial Carcinoma
Brief Title: Aminopterin in Treating Patients With Recurrent or Refractory Endometrial Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Organization: Sanofi (Industry)
Purpose: Treatment
Other Study IDs: CDR0000066974; ILEX-AMT221-A1; ILEX-AMT221; NCI-V99-1531
Record Dates: First submitted 1999-11-01; First posted 2004-08-04 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2000-07

CONDITIONS: Endometrial Cancer
Keywords: recurrent endometrial carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Aminopterin

INTERVENTIONS:
Drug: aminopterin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of aminopterin in treating patients who have refractory or recurrent endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate the antitumor activity of aminopterin in patients with persistent, recurrent, or refractory endometrial carcinoma who have failed prior first line cytotoxic chemotherapy. II. Determine the quantitative and qualitative toxic effects of aminopterin in this patient population. III. Determine the overall patient survival and time to progression of these patients. IV. Assess the pharmacokinetic profile of these patients.

OUTLINE: Patients receive oral aminopterin every 12 hours twice weekly. Treatment continues for up to 15 months in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months until death.

PROJECTED ACCRUAL: A total of 15-25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed persistent, recurrent, or refractory endometrial carcinoma who have failed prior first line chemotherapy Bidimensionally measurable disease by physical exam or medical imaging techniques (sonography acceptable if lesion(s) are clearly defined and measurable in two dimensions) Ascites and pleural effusions are not measurable

PATIENT CHARACTERISTICS: Age: Not specified Performance status: GOG 0-2 Life expectancy: At least 2 months Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Granulocyte count at least 1,500/mm3 Hemoglobin at least 8 g/dL Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) SGOT no greater than 3 times ULN Alkaline phosphatase no greater than 3 times ULN Renal: Creatinine no greater than 2.0 mg/dL Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No significant infection

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy and recovered Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy and recovered Surgery: At least 4 weeks since prior surgery and recovered Other: At least 4 weeks since any prior therapy directed at malignant endometrial tumor(s) At least 4 weeks since prior folate-containing vitamins No concurrent folate-containing vitamins No other concurrent anticancer therapy

Max Age: 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1998-01

CONTACTS AND LOCATIONS:
Overall Officials: David S. Miller, MD, Study Chair — Simmons Cancer Center
Locations (6):
- United States (6):
  - Division of Gynecologic Oncology, St Louis, Missouri
  - East Carolina University School of Medicine, Greenville, North Carolina
  - Gynecologic Oncologists of NE Ohio, Akron, Ohio
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Texas Oncology, P.A., Dallas, Texas
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin